CLINICAL TRIAL: NCT05433350
Title: Pharmacokinetic, Efficacy, Safety, and Tolerability Study of a Single Dose of Acoziborole Under Fasting Conditions in Paediatric Patients From 1 to 14 Years of Age and With g-HAT: a Multicentre, Open-label Study
Brief Title: Pharmacokinetic, Efficacy, Safety and Tolerability Study of a Single Dose of Acoziborole in g-HAT Paediatric Patients
Acronym: OXA005
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNDi-OXA-05-HAT; ACOZI-KIDS (Other Grant/Funding Number: EDCTP: RIA2019PD-2890)
Record Dates: First submitted 2022-06-15; First posted 2022-06-27 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Trypanosomiasis, African; Trypanosoma Brucei Gambiense; Infection; Sleeping Sickness
Keywords: g-HAT; ACOZI-KIDS
MeSH Terms: conditions — Trypanosomiasis, African; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acoziborole (Experimental): Single dose administration
  Two different mode of administration will be used depending on the body weight and on the step of the study:
  * In step 1: 2 tablets of 320 mg (whole) for paediatric patients weighing 30 to 40 kg
  * In step 2 : whole or crushed tablets (1 or 2 tablets depending on the weight) for paediatric patients weighing 10 to 40 kg. Tablets will be crushed for paediatric patients < 6 years old and for paediatric patients ≥ 6 years old who are unable to swallow tablets
  * Initially, recruitment will be limited to paediatric patients weighing 30 to 40 kg who will receive the 2 tablets of 320 mg.
  * Once the PK data from the first six patients have been analysed and the dosing regimen confirmed or adapted, inclusion will resume and be extended to allow enrolment of paediatric patients weighing >10 kg.
  Interventions: Drug: Acoziborole

INTERVENTIONS:
Drug: Acoziborole — Two different mode of administration will be used during the study depending on the body weight and on the step of the study:
  whole tablets of 320 mg dose for paediatric patients weighing 30 to 40 kg in step 1 whole or crushed tablets for paediatric patients weighing 10 to 40 kg in step 2

SUMMARY:
Acoziborole has been studied in an open-label pivotal Phase II/III trial (DNDi-OXA-02-HAT) in the DRC and Guinea. As the numbers of reported cases diminish, resources for surveillance and specialised screening will also taper. This decrease, coupled with the loss of diagnostic skills and disease management expertise, will lead to a weak and less specialised HAT technical environment. The history of g-HAT has shown that outbreaks or re-emergence of the disease have already happened under different circumstances when surveillance was relaxed or simply because the populations at risk live in areas of political instability, limiting access to specialised care. Even with a steady decrease of reported incidence, no model can currently predict that HAT could not re-emerge.

Although g-HAT is predominantly a disease of adults, children are also affected at diverse rates depending on the geographical and behavioural characteristics in the different areas of disease transmission. Hence efforts are needed to develop a paediatric formulation from a new generation of oral HAT treatments.

DETAILED DESCRIPTION:
Human African trypanosomiasis (HAT), or sleeping sickness, is a life-threatening disease transmitted by tsetse flies and caused by a single-celled extracellular parasite that lives free in the bloodstream and other body fluids, including lymph and cerebrospinal fluid (CSF). There are many species of African trypanosomes; however, only two subspecies of the Trypanosoma brucei (T.b.) species are causative of HAT. T.b. gambiense is endemic in West and Central Africa and causes over 98% of current cases. It progresses at a more indolent pace than that of T.b. rhodesiense.

Approximately 5 million people live in areas, mainly in rural parts of 24 disease endemic countries in West and Central Africa, where HAT due to T.b. gambiense (g-HAT) is still considered a public health problem; whereas, 51 million people are estimated to be at risk of infection on the African continent. With 864 cases of g-HAT reported in 2019, the global goal of sustainable disease elimination by 2030, including the interruption of the transmission of g-HAT, is foreseeable. Consistently falling numbers of cases are thanks to efforts from national control programmes, supported by the World Health Organization (WHO), non-governmental organisations, bilateral cooperation, the private sector (including pharmaceutical companies), and philanthropic organisations.

As the numbers of reported cases diminish, resources for surveillance and specialised screening will also taper. This decrease, coupled with the loss of diagnostic skills and disease management expertise, will lead to a weak and less specialised HAT technical environment. The history of g-HAT has shown that outbreaks or re-emergence of the disease have already happened under different circumstances when surveillance was relaxed, e.g. South Sudan and the Democratic Republic of the Congo (DRC) or simply because the populations at risk live in areas of political instability, limiting access to specialised care. Even with a steady decrease of reported incidence, no model can currently predict that HAT could not re-emerge.

Although g-HAT is predominantly a disease of adults, children are also affected at diverse rates depending on the geographical and behavioural characteristics in the different areas of disease transmission. Globally, the WHO Expert Committee on control and surveillance report states: "rates in children are usually less than half of those in adults, reflecting less exposure to flies during daily activities". In data from the Médecins Sans Frontières Database on HAT control projects, out of 684 second stage HAT patients included, 17.5% were children under the age of 15 hence efforts are needed to develop a paediatric formulation from a new generation of oral HAT treatments. The majority of signs and symptoms associated with HAT occur at similar frequencies in paediatric patients with first and second stage disease compared with adults, including sleep disturbances. The presence of trypanosomes in cervical lymph nodes is less frequent in preschool children than in older children and adults. More infants are seen at the second stage, most likely due to delayed diagnosis and the immaturity of the blood-brain barrier. In some studies, fever, hepatomegaly, splenomegaly and facial oedema were observed more frequently in children aged 2 to 15 years than in adults.

As per the WHO 2019 interim guidelines for the treatment of HAT, the choice treatment is determined by a two-step assessment. The first step is the clinical assessment and the second step is the CSF examination (lumbar puncture), which is required only for patients with clinical symptoms and signs suggestive of the severe meningo-encephalitic stage.

For children <6 years old and <20 kg body weight who are second stage g-HAT, a 7-day, twice a day intravenous course of NECT or eflornithine is the sole treatment option. Treatment in first stage g-Hat involves intramuscular injections of pentamidine for 7 days. Both treatments require pre-treatment lumbar puncture and hospitalisation with a specialised health care environment that is not always possible in remote rural African areas where g-HAT is prevalent.

The aim of the current study is to validate the weight-based exposure based on the population pharmacokinetic (pop-PK) modelling, efficacy, and safety of acoziborole in first and second stage g-HAT paediatric patients from 1 to 14 years of age enabling a paradigm shift in the management of paediatric g-HAT patients reducing the subsequent burden on families (i.e. mothers and the entire family will spend less time providing care). Furthermore, if the clinical status permits, administering a single-dose oral drug at the point of diagnosis will avoid the need for costly hospitalisation in specialised health centres, lumbar puncture and parenteral treatments. Compliance and adherence of children to treatment will be more straightforward and will shorten the delay between diagnosis and effective treatment, which will contribute to stopping disease progression and the avoidance of neurological sequelae in this population.

Achieving the challenging objective of g-HAT elimination by 2030 requires a safe, effective, and easy-to-use tool that enables treatment at the point-of-diagnosis for all individuals, including children. As a single administration oral drug, acoziborole would facilitate treatment access for children.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from one parent or from the legal representative
* Assent from the paediatric patient (for paediatric patients >6 years of age) to participate in the study, collected in the presence of an impartial witness
* Between 1 and 14 years of age and between 10 and ≤40 kg (as per the requirements of step 1 and step 2)
* Male or female
* Evidence of trypanosomes in any body fluid (blood or lymph or CSF)
* Having a permanent address and able to comply with the schedule of follow-up visits
* Agreement to not take part in any other clinical trials during the participation in this study
* For pubescent girls of childbearing potential must agree to have avoid getting pregnant during the screening period and up to 3 months after acoziborole dosing by using an acceptable effective contraception method (sexual abstinence, condom, injectable progestin-only contraceptive)
* Agreement not to continue any treatment (including traditional/herbal medicine) without consulting the investigator
* Agreement not to start a treatment (including traditional/herbal medicine) during 4 months after intake of acoziborole without consulting the Investigator

Exclusion Criteria:

* Previous treatment for g-HAT
* Refusal to participate in the study, expressed by the paediatric patient and/or parent or legal representative
* Complicated severe acute malnutrition as defined by weight for height (-3 SDs Z score)
* Unable to take medication by the oral route
* Clinically significant medical condition (other than HAT) that could, in the opinion of the Investigator, jeopardise the patient's safety or interfere with participation in the study
* Any condition (excluding HAT-specific symptoms) that affects the patient's and/or parent's ability to communicate with the Investigator as required to complete the study
* Prior enrolment in the study or prior intake of acoziborole
* Foreseeable difficulty complying with follow-up, including family of migrant workers, refugee status, itinerant trader, etc.
* Clinically significant laboratory test abnormality, with:

  * Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) more than twice the upper limit of normal (ULN)
  * Total bilirubin more than 1.5 x ULN
  * Severe leukopenia at <2000/mm3
  * Potassium <3.5 mmol/L
  * Any other clinically significant laboratory test abnormality
* Pregnancy confirmed by a positive urine pregnancy test (during the screening period and/or within 24 hours prior to the start of treatment) for pubescent girls of childbearing potential
* Not tested for malaria and/or not having received appropriate treatment for malaria
* Not having received appropriate treatment for soil-transmitted helminthiasis
* Paediatric patient who is taking praziquantel, erythromycin, ritonavir, lopinavir, or darunavir and could not stop this treatment

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2022-07-09 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | From time 0 to 96 hours
  Primary PK parameters in blood
Area under the curve (AUC0-96h) | From time 0 to 96 hours
  Primary PK parameters in blood
Time to maximum concentration (Tmax) | From time 0 to 96 hours
  Primary PK parameters in blood
Area under curve (AUC0-∞) | Day 1 Hour 0, Day 1 Hour 4, Day 1 Hour 9, Day 2 Hour 24, Day 3 Hour 48, Day 4 Hour 72, Day 5 Hour 96, Day 11 Hour 264, month 3 any time
  Secondary PK parameters in blood
Clearance | Day 1 Hour 0, Day 1 Hour 4, Day 1 Hour 9, Day 2 Hour 24, Day 3 Hour 48, Day 4 Hour 72, Day 5 Hour 96, Day 11 Hour 264, month 3 any time
  Secondary PK parameters in blood
Volume of distribution (Vd) | Day 1 Hour 0, Day 1 Hour 4, Day 1 Hour 9, Day 2 Hour 24, Day 3 Hour 48, Day 4 Hour 72, Day 5 Hour 96, Day 11 Hour 264, month 3 any time
  Secondary PK parameters in blood
Half-life (t1/2) | Day 1 Hour 0, Day 1 Hour 4, Day 1 Hour 9, Day 2 Hour 24, Day 3 Hour 48, Day 4 Hour 72, Day 5 Hour 96, Day 11 Hour 264, month 3 any time
  Secondary PK parameters in blood
CSF concentration | Day 11
  Acoziborole concentration in CSF

SECONDARY OUTCOMES:
Success or failure | 6 and 12 months post-treatment
  Assess efficacy of acoziborole. Failure defined as death, if rescue medication is required, if evidence of trypanosome in any body fluid, if WBC in CSF >20 cells, clinical signs or symptoms evoking a failure, lost to follow-up, if post treatment LPs refused
Cumulative risk of proven failure over time (Kaplan-Meyer estimate) | 6 and 12 months post-treatment
  Assess efficacy of acoziborole. Failure defined as death, if rescue medication is required, if evidence of trypanosome in any body fluid, if WBC in CSF >20 cells, clinical signs or symptoms evoking a failure, lost to follow-up, if post treatment LPs refused
Occurrence of any treatment-emergent adverse events (TEAEs) (any grade) during the observation period | Day 1 to month 6
  Assess the safety profile of acoziborole
Occurrence of any TEAEs (grade ≥3 or severe) and relatedness to medication during the observation period | Day 1 to month 6
  Assess the safety profile of acoziborole
Occurrence of any serious adverse events (SAEs) during the study | Day 1 to month 12
  Assess the safety profile of acoziborole
Corrected QT interval (QTc) | Day 1 Hour 0, Day 1 Hour 4, Day 1 Hour 9, Day 2 Hour 24, Day 3 Hour 48, Day 4 Hour 72, Day 5 Hour 96, Day 11 Hour 264
  Assess the potential relationship between concentration of acoziborole and corrected QT interval (QTc)
Palatability questionnaire | Day 1
  Assess the palatability of the paediatric formulation in paediatric patients (only in step 2), questionnaire to be completed by the patient. Scores of the 5-point hedonic scale
Acceptability questionnaire | Day 1
  Assess the acceptability of the paediatric formulation in paediatric patients (only in step 2), questionnaire to be completed by the caregiver. Scores of the 5-point hedonic scale

CONTACTS AND LOCATIONS:
Overall Officials: Victor Kande Betu Ku Mesu, Dr, Principal Investigator — Ministry of Public Health, Hygiene and Prevention, Kinshasa
Locations (6):
- Democratic Republic of the Congo (5):
  - General Hospital of Bandundu, Bandundu Province, Bandundu
  - CDTC Katanda, Katanda, East Kasai
  - Hôpital Général de Dipumba, Mbuji-Mayi, East Kasai
  - HGR Bagata, Bagata, Kwilu
  - Hospital of Masi-Manimba, Masi-Manimba, Kwilu
- General Referral Hospital of Dubreka, Dubréka, Guinea

REFERENCES:
- See also: ACOZI-KIDS project on DNDi website — https://dndi.org/global-networks/acozi-kids/